CLINICAL TRIAL: NCT01935479
Title: A Phase I Study of AK159 in Healthy Postmenopausal Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Asahi Kasei Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: AK159 I-4
Record Dates: First submitted 2013-08-29; First posted 2013-09-05 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2013-09

CONDITIONS: Osteoporosis
Keywords: AK159, teriparatide acetate
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (11):
- AK159 SD 1 (Experimental): Single administration of AK159 dose level 1
  Interventions: Drug: AK159
- AK159 SD 2 (Experimental): Single administration of AK159 dose level 2
  Interventions: Drug: AK159
- AK159 SD 3 (Experimental): Single administration of AK159 dose level 3
  Interventions: Drug: AK159
- AK159 SD 4 (Experimental): Single administration of AK159 dose level 4
  Interventions: Drug: AK159
- MN-10-T SD (Active Comparator): Single administration of teriparatide acetate
  Interventions: Drug: MN-10-T
- AK159 MD 1 (Experimental): Multiple administration of AK159 dose level 1
  Interventions: Drug: AK159
- AK159 MD 2 (Experimental): Multiple administration of AK159 dose level 2
  Interventions: Drug: AK159
- AK159 MD 3 (Experimental): Multiple administration of AK159 dose level 3
  Interventions: Drug: AK159
- AK159 MD 4 (Experimental): Multiple administration of AK159 dose level 4
  Interventions: Drug: AK159
- MN-10-T MD (Active Comparator): Multiple administration of MN-10-T
  Interventions: Drug: MN-10-T
- Placebo MD (Placebo Comparator): Multiple administration of placebo AK159
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AK159 — transdermal administration of teriparatide acetate
  Arms: AK159 MD 1; AK159 MD 2; AK159 MD 3; AK159 MD 4; AK159 SD 1; AK159 SD 2; AK159 SD 3; AK159 SD 4
Drug: MN-10-T — subcutaneous administration of teriparatide acetate
  Arms: MN-10-T MD; MN-10-T SD
Drug: Placebo — Placebo AK159
  Arms: Placebo MD

SUMMARY:
The objective of this study is to investigate the pharmacokinetics, safety, and tolerability of AK159 administered to healthy postmenopausal women.

DETAILED DESCRIPTION:
This study consists of two parts: Part 1 and Part 2. The Part 1 is a single-center, randomized, 2-way crossover study that investigates the pharmacokinetics, safety, and tolerability of teriparatide after a single dose of AK159 (5 levels) and estimates the relative bioavailability of AK159 with subcutaneous teriparatide acetate in healthy post-menopausal women.

The Part 2 is a multiple-center, randomized, double-blind, positive- and placebo-controlled, parallel study that compares the pharmacokinetics, bone makers, safety, and tolerability of teriparatide after a weekly doses of AK159 (4 levels) for 6 weeks with placebo and a weekly doses of subcutaneous teriparatide acetate in healthy post-menopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Healthy postmenopausal ethnic Japanese women
* At least 45 years of age at the time consent is obtained
* Give voluntary consent in writing with a sufficient understanding of the study.

Exclusion Criteria:

* Clinical abnormality identified in the laboratory tests
* Weight < 40.0 kg
* Body mass index < 17.5 or >=30.5
* History of disease of the kidneys, liver, heart, brain, or other organ that makes them ineligible as subjects
* Previously received radiation treatment potentially affecting bone
* Clinical abnormality identified in the 12-lead ECGs performed at the study center during the screening period
* Systolic blood pressure < 90 mmHg
* Serum calcium level exceeding 10.4 mg/dL
* History of contact dermatitis or skin disease potentially compromising study evaluation
* Used drugs which impact bone metabolism in the 8-week period preceding investigational product administration
* Used a bisphosphonate
* Used a teriparatide product

Min Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of teriparatide | up to 6 hours after single and repeated administration
Peak Plasma Concentration (Cmax) of teriparatide | up to 6 hours after single and repeated administration
Number of subjects with adverse events and Incidence of adverse events | up to 7 weeks after the initial administration
Change in bone turnover markers from baseline | up to 7 weeks after the initial administration

SECONDARY OUTCOMES:
Visual assessment of the application site | up to 7 weeks after the initial administration

OTHER OUTCOMES:
Residual teriparatide in the patch after application | up to 6 weeks after the initial administration

CONTACTS AND LOCATIONS:
Locations (3):
- Japan (3):
  - Fukuoka
  - Kumamoto
  - Sumida City